CLINICAL TRIAL: NCT00592124
Title: Phase 2 Adherence and Pharmacokinetics Study of Oral and Vaginal Preparations of Tenofovir
Brief Title: Adherence and Acceptability to and Blood Levels of Tenofovir Gel and Tablets in HIV Uninfected Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Microbicide Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MTN-001; 10617 (Registry Identifier: DAIDS ES); 1U01AI068633-01 (NIH)
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: Microbicide; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): Oral tenofovir disoproxil fumarate (TDF) for Weeks 1 through 6, vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF and vaginal tenofovir gel application for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel
- 2 (Experimental): Vaginal tenofovir gel application for Weeks 1 through 6, oral TDF for Weeks 8 through 13, and oral TDF and vaginal tenofovir gel application for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel
- 3 (Experimental): Oral TDF and vaginal tenofovir gel application for Weeks 1 through 6, oral TDF for Weeks 8 through 13, and vaginal tenofovir gel application for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel
- 4 (Experimental): Oral TDF and vaginal tenofovir gel application for Weeks 1 through 6, vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel
- 5 (Experimental): Oral TDF for Weeks 1 through 6, oral TDF and vaginal tenofovir gel application for Weeks 8 through 13, and vaginal tenofovir gel application for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel
- 6 (Experimental): Vaginal tenofovir gel application for Weeks 1 through 6, oral TDF and vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF for Weeks 15 through 20
  Interventions: Drug: Tenofovir disoproxil fumarate; Drug: Tenofovir gel

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate — 300 mg tablet daily
  Other Names: TDF
Drug: Tenofovir gel — 1 gm/100 ml of 1% gel vaginally daily
  Other Names: TFV; 9-[2-(Phosphonomethoxy)propyl]adenine

SUMMARY:
A new approach to HIV prevention currently being studied includes the use of microbicides, substances that kill microbes. Tenofovir disoproxil fumarate (TDF) is an oral, FDA-approved, anti-HIV drug, and tenofovir gel is an experimental microbicide. The purpose of this study is to determine the adherence and acceptability to and blood levels of three daily regimens of tenofovir in both oral and gel form.

DETAILED DESCRIPTION:
It is necessary to monitor both the adherence and blood levels of microbicides in order to gauge its efficacy in a study population. Utilizing an experimental microbicide (tenofovir gel) and an anti-HIV drug (TDF), this study will measure the adherence and acceptability to and blood levels of the two interventions in three separate regimens given to HIV-uninfected women.

The expected duration of participation for each participant is 21 weeks. Study participants will be randomly assigned into one of six study groups, each with a different regimen sequence. Each sequence will consist of three study periods and three wash-out periods. Each study period lasts 6 weeks, followed by a 1 week wash-out period. The regimen assigned for a given study period will include either oral TDF, tenofovir vaginal gel, or both. All participants will be prescribed all three regimens in the order designated by their randomized assignment.

Study visits will occur at Weeks 1, 3, 6, 7, 10, 13, 14, 17, 20, and 21. Medical history, a physical exam, behavioral assessment, and urine, blood, pelvic sample collection, and counseling will occur at all visits. At some study sites rectal swabs may be performed. Counseling will include information regarding contraception, protocol adherence, HIV, HIV/Sexually Transmitted Infection risk reduction, and male condom use. Pharmacokinetic (PK) studies, to be determined by the study site, will occur during all three study periods. These studies may involve additional procedures.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* HIV-uninfected
* Normal menstrual cycle. More information can be found in the protocol.
* Creatinine clearance greater than 70 ml/min
* Sexually active. More information can be found in the protocol.
* Normal Pap smear result within 12 months prior to study entry
* Agrees to not participate in other investigational studies
* Willing to use effective forms of contraception. More information can be found in the protocol.

Exclusion Criteria:

* Adverse reaction to either of the study products
* Adverse reaction to latex
* Currently sexually active with a partner with history of adverse reaction to latex
* More than three sexual partners in the month prior to screening
* Pathologic bone fracture not related to trauma
* Last pregnancy outcome within 90 days or less prior to enrollment
* Gynecologic or genital procedure within 90 days of study entry
* Enrollment in other investigational study within 30 days of study entry
* Nontherapeutic injection drug use within 12 months of screening
* Any social or medical condition that, in the opinion of the investigator, would interfere with the study
* Abnormal laboratory values
* Grade 2 or higher genital lesions, erythema, and/or edema or has any other abnormal physical or pelvic exam finding that, in the opinion of the investigator, would interfere with the study
* Kidney, reproductive, or urinary tract infection requiring treatment. More information on this criterion can be found in the protocol.
* Pregnant, breastfeeding, or intend to become pregnant
* Unwilling to comply with study participation requirements, including attendance at all scheduled study visits
* Per participant report, use of the following at enrollment, and/or anticipated use during the period of study participation - use of a diaphragm, vaginal ring, and/or spermicide for contraception, acyclovir or valacyclovir, post-exposure prophylaxis for HIV exposure, TDF/emtricitabine, non-study vaginal products

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig W. Hendrix, MD, Study Chair — Johns Hopkins University
Locations (7):
- United States (4):
  - Alabama Microbicide CRS, Birmingham, Alabama
  - Bronx- Lebanon Hospital Center Clinical Research Site (BLHC CRS), The Bronx, New York
  - Case CRS, Cleveland, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
- South Africa (2):
  - Botha's Hill CRS, Durban, KwaZulu-Natal
  - Umkomaas CRS, Durban, KwaZulu-Natal
- Makerere University- JHU Research Collaboration {MUJHU CARE LTD} CRS, Kampala, Uganda

REFERENCES:
- [Background] Bateman C. Tenofovir gel--the new HIV prevention 'banker'? S Afr Med J. 2007 Jul;97(7):496, 498. No abstract available. PMID 17805450
- [Background] Mayer KH, Maslankowski LA, Gai F, El-Sadr WM, Justman J, Kwiecien A, Masse B, Eshleman SH, Hendrix C, Morrow K, Rooney JF, Soto-Torres L; HPTN 050 Protocol Team. Safety and tolerability of tenofovir vaginal gel in abstinent and sexually active HIV-infected and uninfected women. AIDS. 2006 Feb 28;20(4):543-51. doi: 10.1097/01.aids.0000210608.70762.c3. PMID 16470118
- [Result] Hendrix CW, Chen BA, Guddera V, Hoesley C, Justman J, Nakabiito C, Salata R, Soto-Torres L, Patterson K, Minnis AM, Gandham S, Gomez K, Richardson BA, Bumpus NN. MTN-001: randomized pharmacokinetic cross-over study comparing tenofovir vaginal gel and oral tablets in vaginal tissue and other compartments. PLoS One. 2013;8(1):e55013. doi: 10.1371/journal.pone.0055013. Epub 2013 Jan 30. PMID 23383037
- [Derived] Minnis AM, van der Straten A, Salee P, Hendrix CW. Pre-exposure Prophylaxis Adherence Measured by Plasma Drug Level in MTN-001: Comparison Between Vaginal Gel and Oral Tablets in Two Geographic Regions. AIDS Behav. 2016 Jul;20(7):1541-8. doi: 10.1007/s10461-015-1081-3. PMID 25969178
- [Derived] Minnis AM, Gandham S, Richardson BA, Guddera V, Chen BA, Salata R, Nakabiito C, Hoesley C, Justman J, Soto-Torres L, Patterson K, Gomez K, Hendrix CW. Adherence and acceptability in MTN 001: a randomized cross-over trial of daily oral and topical tenofovir for HIV prevention in women. AIDS Behav. 2013 Feb;17(2):737-47. doi: 10.1007/s10461-012-0333-8. PMID 23065145

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in this study were selected from a total of 7 multinational clinical research sites, with first enrollment taking place on 4 March 2009 and last on 3 February 2010.
Groups:
- O, V, OV: Oral tenofovir disoproxil fumarate (TDF) for Weeks 1 through 6, vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF and vaginal tenofovir gel application for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
- V, O, OV: Vaginal tenofovir gel application for Weeks 1 through 6, oral TDF for Weeks 8 through 13, and oral TDF and vaginal tenofovir gel application for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
- OV, O, V: Oral TDF and vaginal tenofovir gel application for Weeks 1 through 6, oral TDF for Weeks 8 through 13, and vaginal tenofovir gel application for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
- OV, V, O: Oral TDF and vaginal tenofovir gel application for Weeks 1 through 6, vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
- O, OV, V: Oral TDF for Weeks 1 through 6, oral TDF and vaginal tenofovir gel application for Weeks 8 through 13, and vaginal tenofovir gel application for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
- V, OV, O: Vaginal tenofovir gel application for Weeks 1 through 6, oral TDF and vaginal tenofovir gel application for Weeks 8 through 13, and oral TDF for Weeks 15 through 20
  Tenofovir disoproxil fumarate: 300 mg tablet daily
  Tenofovir gel: 1 gm/100 ml of 1% gel vaginally daily
Period: Overall Study
Arm/Group | O, V, OV | V, O, OV | OV, O, V | OV, V, O | O, OV, V | V, OV, O
Started | 28 | 29 | 30 | 27 | 27 | 27
Completed | 24 | 24 | 24 | 24 | 24 | 24
Not Completed | 4 | 5 | 6 | 3 | 3 | 3

BASELINE CHARACTERISTICS:
Population: The baseline population consists of evaluable enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | O, V, OV | V, O, OV | OV, O, V | OV, V, O | O, OV, V | V, OV, O | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (7.6) | 29.1 (6.3) | 29.8 (6.5) | 31.3 (6.4) | 31.1 (7.5) | 31.3 (8.2) | 30.8 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 24 | 24 | 24 | 24 | 144
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 0 | 2 | 0 | 1 | 6
  Not Hispanic or Latino | 11 | 10 | 12 | 10 | 13 | 11 | 67
  Unknown or Not Reported | 12 | 12 | 12 | 12 | 11 | 12 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race categories applicable to USA participants only.
  Participants
    number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 72
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Asian | 0 | 2 | 0 | 1 | 0 | 0 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 7 | 4 | 9 | 4 | 6 | 5 | 35
    White | 5 | 6 | 3 | 6 | 5 | 7 | 32
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 12 | 72
  South Africa | 8 | 8 | 8 | 8 | 8 | 8 | 48
  Uganda | 4 | 4 | 4 | 4 | 4 | 4 | 24
Are you currently married? [Count of Participants; unit: Participants]
  Yes | 9 | 9 | 8 | 10 | 9 | 12 | 57
  No | 15 | 15 | 16 | 14 | 15 | 12 | 87
Do you currently have a male sex partner? [Count of Participants; unit: Participants]
  Yes | 15 | 15 | 16 | 13 | 14 | 12 | 85
  No | 9 | 9 | 8 | 11 | 10 | 12 | 59
What is your household(s) average monthly income? [Median (Inter-Quartile Range); unit: US Dollars] — Population: Four participants did not provide information on household income.
  US Dollars
    number analyzed (Participants) | 24 | 23 | 24 | 23 | 23 | 23 | 140
    (all) | 495.40 [227.00 to 1250.00] | 773.01 [122.70 to 3200.00] | 417.18 [141.75 to 940.80] | 490.80 [147.24 to 2400.00] | 368.10 [98.16 to 1500.00] | 306.75 [98.16 to 2500.00] | 495.40 [134.99 to 1900.00]
What is your highest education level? [Count of Participants; unit: Participants]
  No Schooling | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Primary School, Not Complete | 1 | 3 | 1 | 2 | 0 | 1 | 8
  Primary School, Complete | 0 | 1 | 2 | 1 | 1 | 2 | 7
  Secondary School, Not Complete | 7 | 5 | 4 | 6 | 7 | 8 | 37
  Secondary School, Complete | 8 | 3 | 6 | 4 | 6 | 2 | 29
  Attended College or University | 8 | 12 | 11 | 11 | 9 | 11 | 62

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Adherence to Each Regimen
Description: Participant self-reported product use. For each woman, adherence to each regimen was computed by dividing the number of daily doses she reported having taken by the number of doses expect if she were fully adherent.
Time Frame: Measured through Week 21
Population: For each woman, adherence to each regimen was computed by dividing the number of daily doses she reported having taken by the number of expected doses if she were fully adherent.
Measure: Mean (Standard Deviation); unit: percentage of expected doses
Groups:
- Vaginal and Oral Tenofovir: TDF 300 mg tablet (oral tenofovir) and tenofovir 1% gel (vaginal tenofovir)
- Oral Tenofovir: TDF 300 mg tablet (oral tenofovir)
- Vaginal Tenofovir: Tenofovir 1% gel (vaginal tenofovir)
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
percentage of expected doses | 94 (10.8) | 93.8 (10.2) | 93.9 (10.1)

2. Primary Outcome: Proportion of Participants Who Indicate They Would be "Unlikely" Use Study Product in the Future
Time Frame: Measured through Week 21
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 141 | 139 | 142
Participants
  Likely | 115 | 130 | 117
  Unlikely | 26 | 9 | 25

3. Primary Outcome: Systemic and Local PK Among Three Regimens of Tenofovir (Oral, Vaignal, and Dual Use)
Description: PK measures, including maximum concentrations (Cmax) in serum, tissue, and cervicovaginal lavage.
Time Frame: Measured through Week 21
Population: Serum TFV and Tissue TFV measures do not include participants from South Africa clinical sites.
Measure: Median (Inter-Quartile Range); unit: ng/mL, ng/mg, ng/mL
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
ng/mL, ng/mg, ng/mL
  Serum TFV Cmax: number analyzed (Participants) | 128 | 128 | 128
  Serum TFV Cmax | 337 [257 to 447] | 332 [257 to 406] | 3.9 [2.2 to 7.9]
  Tissue TFV: number analyzed (Participants) | 128 | 128 | 128
  Tissue TFV | 104 [40 to 268] | 0.15 [0.15 to 0.20] | 113 [27 to 265]
  Cervicovaginal lavage | 1600000 [500000 to 6500000] | 5380 [6 to 201560] | 3100000 [600000 to 8100000]

4. Secondary Outcome: Frequency of Product Use
Description: This number represents how often participant used study product during the preceding 3 weeks and is measured twice during each 6 week product period.
Time Frame: Measured through Week 21
Measure: Count of Units; unit: 3-week periods
Units Other Than Participants: 3-week periods
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
Number analyzed (3-week periods) | 283 | 282 | 285
3-week periods
  Never | 0 | 1 | 3
  Less than once/week | 1 | 1 | 0
  1-3 times/week | 7 | 5 | 9
  4-6 times/week | 48 | 59 | 41
  Once/day | 227 | 216 | 232

5. Secondary Outcome: Number of Days Product Missed
Description: This represents the longest number of days in a row during the past 3 weeks that a participant missed using the study product.
Time Frame: Measured through Week 21
Population: This outcome is based on evaluable participants.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: 3-week periods
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
Number analyzed (3-week periods) | 283 | 282 | 284
days | 0.9 (1.9) | 0.9 (2.3) | 0.9 (2.4)

6. Secondary Outcome: Proportion of Women Who Report Taking at Least 90% of Expected Daily Doses
Time Frame: Measured through Week 21
Population: This outcome is based on evaluable participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
Participants
  Yes | 114 | 114 | 122
  No | 30 | 30 | 22

7. Secondary Outcome: Frequency of Sexual Activity
Description: This represents the rate during the past 3 weeks at which participants engaged in vaginal sex.
Time Frame: Measured through Week 21
Measure: Count of Units; unit: 3-week periods
Units Other Than Participants: 3-week periods
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
Number analyzed (3-week periods) | 264 | 272 | 271
3-week periods
  Less than once/week | 18 | 14 | 10
  1-3 times/week | 170 | 179 | 184
  4-6 times/week | 58 | 55 | 48
  Once/day | 11 | 18 | 17
  More than once/day | 7 | 6 | 12

8. Secondary Outcome: Frequency of Male Condom Use
Time Frame: Measured through Week 21
Measure: Count of Units; unit: 3-week periods
Units Other Than Participants: 3-week periods
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144 | 144
Number analyzed (3-week periods) | 266 | 272 | 271
3-week periods
  Never | 71 | 80 | 69
  Rarely | 19 | 21 | 28
  Sometimes | 22 | 24 | 15
  Most of the time | 26 | 27 | 28
  Always | 128 | 120 | 131

9. Secondary Outcome: Tablet Usage Before Sex
Description: These summaries represent counts and percentages of participants using tablet before last instance of vaginal sex.
Time Frame: Measured through Week 21
Population: Last instance of vaginal intercourse on the same day as tablet use
Measure: Count of Units; unit: Sexual encounters
Units Other Than Participants: Sexual encounters
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual encounters) | 254 | 266
Sexual encounters
  Yes | 150 | 186
  No | 104 | 80

10. Secondary Outcome: Length of Time Vaginal Sexual Intercourse Took Place After Using Tablet.
Description: Median and inter-quartile range of the time between product usage and instance of vaginal intercourse (given tablet was used before the encounter).
Time Frame: Measured through Week 21
Population: Last instances of vaginal sexual intercourse wherein tablets were used before the encounters. Timing data was not provided for four sexual encounters.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 148 | 184
minutes | 60.0 [45.0 to 180.0] | 90.0 [60.0 to 180.0]

11. Secondary Outcome: Tablet Usage After Sex
Description: These summaries represent counts and percentages of participants using tablet after last instance of vaginal sex.
Time Frame: Measured through Week 21
Population: Last instance of vaginal intercourse on the same day as tablet use
Measure: Count of Units; unit: Sexual Encounters
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 255 | 266
Sexual Encounters
  Yes | 105 | 83
  No | 150 | 183

12. Secondary Outcome: Length of Time Vaginal Sexual Intercourse Took Place Before Using Tablet.
Description: Median and inter-quartile range of the time between product usage and instance of vaginal intercourse (given tablet was used after the encounter).
Time Frame: Measured through Week 21
Population: Last instances of vaginal sexual intercourse wherein tablets were used after the encounters. Timing data was not provided for two sexual encounters.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 103 | 83
minutes | 90.0 [45.0 to 180.0] | 120.0 [60.0 to 240.0]

13. Secondary Outcome: Gel Usage Before Sex
Description: These summaries represent counts and percentages of participants using gel before last instance of vaginal sex.
Time Frame: Measured through Week 21
Population: Last instance of vaginal intercourse on the same day as gel use
Measure: Count of Units; unit: Sexual Encounters
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 253 | 262
Sexual Encounters
  Yes | 142 | 151
  No | 111 | 111

14. Secondary Outcome: Length of Time Vaginal Sexual Intercourse Took Place After Using Gel.
Description: Median and inter-quartile range of the time between product usage and instance of vaginal intercourse (given gel was used before the encounter).
Time Frame: Measured through Week 21
Population: Last instances of vaginal sexual intercourse wherein gel was used before the encounters.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 142 | 151
minutes | 60.0 [30.0 to 180.0] | 60.0 [30.0 to 180.0]

15. Secondary Outcome: Gel Usage After Sex
Description: These summaries represent counts and percentages of participants using gel after last instance of vaginal sex.
Time Frame: Measured through Week 21
Population: Last instance of vaginal intercourse on the same day as gel use
Measure: Count of Units; unit: Sexual Encounters
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 254 | 261
Sexual Encounters
  Yes | 112 | 114
  No | 142 | 147

16. Secondary Outcome: Length of Time Vaginal Sexual Intercourse Took Place Before Using Gel.
Description: Median and inter-quartile range of the time between product usage and instance of vaginal intercourse (given gel was used after the encounter).
Time Frame: Measured through Week 21
Population: Last instances of vaginal sexual intercourse wherein gel was used after the encounters.
Measure: Median (Inter-Quartile Range); unit: minutes
Units Other Than Participants: Sexual Encounters
Arm/Group | Vaginal and Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 144 | 144
Number analyzed (Sexual Encounters) | 112 | 114
minutes | 75.0 [52.5 to 180.0] | 120.0 [60.0 to 240.0]

17. Secondary Outcome: Reported Sharing of Product
Description: Number and percentage of participants who had a product sharing event during the 6-week product use period, where a sharing event includes 1) being asked for the study product, or 2) selling, trading, or giving away study product, or 3) having someone take the study product from the participant.
Time Frame: Measured through Week 21
Population: Participants who completed a product sharing assessment at the end of the 6-week product use period.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 139 | 142 | 141
Participants | 2 | 0 | 3

18. Secondary Outcome: Grade 3 or Higher Toxicity for Systemic and Local Effects as Defined by the Protocol
Time Frame: Measured through Week 21
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Number analyzed (Participants) | 168 | 168 | 168
Participants | 5 | 5 | 3

ADVERSE EVENTS:
Time Frame: 21 Weeks
Arm/Group | Vaginal and Oral Tenofovir | Oral Tenofovir | Vaginal Tenofovir
Serious Adverse Events (participants affected / at risk) | 1/168 | 3/168 | 1/168
Other Adverse Events (participants affected / at risk) | 86/168 | 89/168 | 64/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaginal and Oral Tenofovir (N=168) | Oral Tenofovir (N=168) | Vaginal Tenofovir (N=168)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Malaria (Infections and infestations) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaginal and Oral Tenofovir (N=168) | Oral Tenofovir (N=168) | Vaginal Tenofovir (N=168)
Diarrhoea (Gastrointestinal disorders) | 10 | 9 | 3
Nausea (Gastrointestinal disorders) | 24 | 25 | 5
Vomiting (Gastrointestinal disorders) | 7 | 12 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 17 | 10
Vulvovaginal candidiasis (Infections and infestations) | 3 | 9 | 2
Blood phosphorus decreased (Investigations) | 5 | 11 | 6
Haemoglobin decreased (Investigations) | 8 | 8 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 26 | 26 | 18
Headache (Nervous system disorders) | 14 | 8 | 3
Vaginal discharge (Reproductive system and breast disorders) | 10 | 13 | 7
Vulvovaginal pruritus (Reproductive system and breast disorders) | 16 | 9 | 13

LIMITATIONS AND CAVEATS:
For a full discussion of the difficulties of sampling and comparing findings in the varied and complex anatomic spaces in this study, please see the primary results publication, listed in the References section (PLoS One 2013;8(1):e55013.)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No